CLINICAL TRIAL: NCT01984788
Title: A Phase 2a Double-Blind Placebo-Controlled 2-Period Crossover Study to Evaluate the Safety and Efficacy of BCX4161 as a Prophylactic Treatment to Reduce the Frequency of Attacks in Subjects With Hereditary Angioedema
Brief Title: Safety and Efficacy of Oral BCX4161 as a Prophylactic Treatment for HAE
Acronym: OPuS-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioCryst Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: BCX4161-203
Record Dates: First submitted 2013-11-05; First posted 2013-11-15 (Estimated); Last update posted 2014-08-18 (Estimated); Status verified 2014-08

CONDITIONS: Hereditary Angioedema
Keywords: Oral Prophylaxis
MeSH Terms: conditions — Angioedemas, Hereditary | interventions — avoralstat

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BCX4161 (Active Comparator): 400 mg TID for 28 days
  Interventions: Drug: BCX4161
- Placebo (Placebo Comparator): TID for 28 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BCX4161
  Arms: BCX4161
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether BCX4161 given as a daily oral prophylactic treatment is safe and effective in reducing the number of acute attacks in patients with hereditary angioedema.

ELIGIBILITY:
Key Inclusion Criteria:

* Written informed consent
* Clinical and laboratory diagnosis of Hereditary Angioedema Type I or II
* An average angioedema attack frequency of 1/week
* Acceptable birth control measures

Key Exclusion Criteria:

* Concurrent use of defined treatments for prophylaxis
* Pregnancy or breast-feeding
* Clinically significant medical condition, laboratory abnormality or medical history

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-11; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Number of acute angioedema attacks | Over 28 days of treatment

SECONDARY OUTCOMES:
Incidence and severity of adverse events and laboratory abnormalities | Over 28 days of treatment
Number of attack free days | Over 28 days of treatment
Angioedema Quality of Life scores | Over 28 days of treatment
Angioedema activity scores | Over 28 days of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Maurer, MD, Principal Investigator — Charite University, Berlin, Germany
Locations (6):
- Germany (5):
  - Dr Marcus Maurer, Berlin
  - Dr Emel Aygoren-Pursun, Frankfurt
  - Dr Petra Staubach, Mainz
  - Dr Inmaculada Martinez-Saguer, Mörfelden-Walldorf
  - Dr Murat Bas, München
- Dr Hilary Longhurst, London, United Kingdom

REFERENCES:
- [Derived] Beard N, Frese M, Smertina E, Mere P, Katelaris C, Mills K. Interventions for the long-term prevention of hereditary angioedema attacks. Cochrane Database Syst Rev. 2022 Nov 3;11(11):CD013403. doi: 10.1002/14651858.CD013403.pub2. PMID 36326435